CLINICAL TRIAL: NCT01420081
Title: A RANDOMIZED PHASE 2 NON-COMPARATIVE STUDY OF THE EFFICACY OF PF-04691502 AND PF-05212384 IN PATIENTS WITH RECURRENT ENDOMETRIAL CANCER
Brief Title: A Study Of Two Dual PI3K/mTOR Inhibitors, PF-04691502 And PF-05212384 In Patients With Recurrent Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1271004; 2011-003062-32 (EudraCT Number)
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Endometrial Neoplasms
Keywords: uterine neoplasms; endometrial; uterine; cancer; PI3K; mTOR; PI3K/mTOR; recurrent; metastatic
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Neoplasms; Recurrence; Neoplasm Metastasis | interventions — gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Experimental): PI3K Basal, IV Compound
  Interventions: Drug: PF-05212384
- C (Experimental): PI3K Activated, Oral Compound
  Interventions: Drug: PF-05212384
- F (Experimental): Japanese lead in cohort, IV compound
  Interventions: Drug: PF-05212384

INTERVENTIONS:
Drug: PF-05212384 — 154mg IV weekly
  Other Names: PKI-587
  Arms: B
Drug: PF-05212384 — 154mg IV weekly
  Other Names: PKI-587
  Arms: C
Drug: PF-05212384 — 154mg IV weekly
  Other Names: PKI-587
  Arms: F

SUMMARY:
This study will investigate the individual safety and efficacy of two dual PI3K/mTOR inhibitors in patients with recurrent endometrial cancer.

DETAILED DESCRIPTION:
The study was prematurely discontinued due to lack confidence in the Stathmin assay as a patient selection criteria and subsequent lack of confidence in the efficacy signal that was observed. The decision to terminate the study was made on January 23, 2014. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent endometrial carcinoma
* Disease progression following one or two lines of prior treatment with platinum containing chemotherapy
* Tumor tissue available at time of screening for PI3K analysis
* Adequate performance status
* Adequate glucose control, bone marrow, kidney, liver, and heart function

Exclusion Criteria:

* More than 2 prior cytotoxic chemo regimens for endometrial carcinoma
* Prior therapy with an agent known to be a PI3K, and or mTOR and or AKT inhibitor
* Active brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2012-01-19 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2015-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, IDS Pharmacy, Birmingham, Alabama
  - University of California Medical Center, La Jolla, California
  - Moores UC San Diego Cancer Center, La Jolla, California
  - University of California Medical Center, San Diego, California
  - Mercy Hospital, Miami, Florida
  - Mercy Research Institute, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Medicine Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - University of Kansas, Fairway, Kansas
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - Mary Bird Perkins Cancer Center at St. Tammany Parish Hospital, Covington, Louisiana
  - Women's Cancer Care, Covington, Louisiana
  - Women's Cancer Care, Metairie, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
- Peter MacCallum Cancer Centre, Division of Cancer Madicine, East Melbourne, Victoria, Australia
- Canada (8):
  - Foothills Medical Center, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
- Japan (4):
  - Aichi cancer center hospital, Nagoya, Aichi-ken
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
- Poland (3):
  - Regionalny Osrodek Onkologiczny Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - Zaklad Radiologii, Lodz
  - Centrum Onkologii Ziemi Lubelskiej im. Św. Jana z Dukli, Lublin
- Russia (4):
  - Federal State Healthcare Institution, Lermontov, Stavropol Territory
  - Clinical Oncology Dispensary 1 of Department of Healthcare of the Krasnodar Region, Krasnodar
  - Pyatigorsk Oncology Center, Pyatigorsk
  - Saint Petersburg State Healthcare Institution City Clinical Oncology Dispensary, Saint Petersburg
- Spain (6):
  - Hospital Universitari Vall d'hebron, Barcelona
  - Centro Oncologico MD Anderson Internacional España, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Fundacion Instituto Valenciano de Oncologia - I.V.O., Valencia
  - Fundacion Instituto Valenciano de Oncologia - I.V.O, Valencia
- United Kingdom (4):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Beatson Oncology Centre, Glasgow
  - University College London Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Del Campo JM, Birrer M, Davis C, Fujiwara K, Gollerkeri A, Gore M, Houk B, Lau S, Poveda A, Gonzalez-Martin A, Muller C, Muro K, Pierce K, Suzuki M, Vermette J, Oza A. A randomized phase II non-comparative study of PF-04691502 and gedatolisib (PF-05212384) in patients with recurrent endometrial cancer. Gynecol Oncol. 2016 Jul;142(1):62-69. doi: 10.1016/j.ygyno.2016.04.019. Epub 2016 Apr 24. PMID 27103175
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1271004&StudyName=A%20Study%20Of%20two%20dual%20PI3K/mTOR%20inhibitors%2C%20PF-04691502%20And%20PF-05212384%20In%20Patients%20With%20Recurrent%20Endometrial%20Cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, Phase 2, four-arm, non-comparative study to assess the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of PF-04691502 (an oral PI3K/mTOR inhibitor) and PF-05212384 (an Intravenous [IV] Phosphoinositide 3-Kinase [PI3K]/Mammalian Target of Rapamycin [mTOR] inhibitor).
Pre-assignment Details: This study was conducted in parallel-arms in adult participants with recurrent endometrial cancer. Randomized arms included PF-05212384 (154mg dosage) and PF-04691502 (8mg which was lowered to 6mg) for both PI3K Basal or Activated. Lead-in Cohorts included PF-05212384 (89mg or 154mg) and PF-04691502 (4mg).
Groups:
- PF-04691502 8 mg (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants self-administered PF-04691502 8 mg orally, once daily (QD) until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death. Dose of the participants were reduced to 6 mg if they were on 8 mg dose.
- PF-04691502 6 mg (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants self-administered PF-04691502 6 mg orally, QD until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- PF-04691502 8 mg (PI3K Activated): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K activated). Participants self-administered PF-04691502 8 mg orally, QD until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death. Dose of the participants were reduced to 6 mg if they were on 8 mg dose.
- PF-04691502 6 mg (PI3K Activated): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K activated). Participants self-administered PF-04691502 6 mg orally, QD until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- PF-05212384 154 mg (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants received PF-05212384 154 mg by 30 minute infusion at the study site, once weekly (Quaque, QW) until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- PF-05212384 154 mg (PI3K Activated): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K activated). Participants received PF-05212384 154 mg by 30 minute infusion at the study site, QW until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- Lead-in-cohort (LIC) PF-04691502 (4 mg): Participants who were enrolled in the PF-04691502 LIC began dosing with PF-04691502 4 mg at least 4 days (but no more than 10 days) prior to Cycle 1 Day 1 and continued taking PF-05691502 until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- LIC PF-05212384 (89 mg): Participants who were enrolled in the PF-05212384 LIC began dosing with PF-05212384 89 mg at least 4 days (but no more than 10 days) prior to Cycle 1 Day 1 and continued taking PF-05212384 until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- LIC PF-05212384 (154 mg): Participants who were enrolled in the PF-05212384 LIC began dosing with PF-05212384 154 mg at least 4 days (but no more than 10 days) prior to Cycle 1 Day 1 and continued taking PF-05212384 until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
Period: Overall Study
Arm/Group | PF-04691502 8 mg (PI3K Basal) | PF-04691502 6 mg (PI3K Basal) | PF-04691502 8 mg (PI3K Activated) | PF-04691502 6 mg (PI3K Activated) | PF-05212384 154 mg (PI3K Basal) | PF-05212384 154 mg (PI3K Activated) | Lead-in-cohort (LIC) PF-04691502 (4 mg) | LIC PF-05212384 (89 mg) | LIC PF-05212384 (154 mg)
Started | 3 | 1 | 11 | 3 | 20 | 20 | 3 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 11 | 3 | 20 | 20 | 3 | 3 | 3
Not completed — Death | 1 | 0 | 8 | 0 | 7 | 12 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 1 | 1 | 3 | 11 | 7 | 3 | 2 | 2
Not completed — Subject Refused Futher Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-04691502 8 mg (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants self-administered PF-04691502 8 mg orally, QD until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death. Dose of the participants were reduced to 6 mg if they were on 8 mg dose.
- PF-05212384 154 mg (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants received PF-05212384 154 mg by 30 minute infusion at the study site, QW until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- Total: Total of all reporting groups
Arm/Group | PF-04691502 8 mg (PI3K Basal) | PF-04691502 6 mg (PI3K Basal) | PF-04691502 8 mg (PI3K Activated) | PF-04691502 6 mg (PI3K Activated) | PF-05212384 154 mg (PI3K Basal) | PF-05212384 154 mg (PI3K Activated) | Lead-in-cohort (LIC) PF-04691502 (4 mg) | LIC PF-05212384 (89 mg) | LIC PF-05212384 (154 mg) | Total
Number analyzed (Participants) | 3 | 1 | 11 | 3 | 20 | 20 | 3 | 3 | 3 | 67
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 44 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  45 - 64 years | 2 | 1 | 4 | 3 | 9 | 4 | 2 | 1 | 2 | 28
  >= 65 years | 1 | 0 | 7 | 0 | 11 | 16 | 1 | 1 | 1 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 11 | 3 | 20 | 20 | 3 | 3 | 3 | 67
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Response for PF-04691502
Description: Clinical benefit response was defined as best overall response of complete response (CR), partial response (PR) or stable disease (SD) for at least 16 weeks from Cycle 1 Day 1 (C1D1) to the first time of disease progression. The outcome data table below presents the number of participants with clinical benefit response as "yes" or "no". On 09 Oct 2012, Pfizer decided to stop enrollment into PF-04691502. While tumor assessment for PF-04691502 was included as a listing in the final report, formal efficacy analysis for PF-04691502 was not performed.
Time Frame: 16 weeks from Cycle 1 Day 1
Population: Per protocol dataset included participants enrolled for treatment, with baseline tumor, measurable disease and with disease under study. The LIC reporting arm were not a part of the per protocol analysis set for summarizing response.
Measure: Number; unit: Participants
Groups:
- PF-04691502 (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants self-administered PF-04691502 orally, QD until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
- PF-04691502 (PI3K Activated): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K activated). Participants self-administered PF-04691502 orally, QD until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
Arm/Group | PF-04691502 (PI3K Basal) | PF-04691502 (PI3K Activated)
Number analyzed (Participants) | 4 | 11
Participants
  Participants with "Yes" response | 1 | 0
  Participants with "No" response | 3 | 11

2. Primary Outcome: Percentage of Participants With Clinical Benefit Response for PF-05212384
Description: Clinical benefit response was defined as best overall response of complete response (CR), partial response (PR) or stable disease (SD) for at least 16 weeks from Cycle 1 Day 1 (C1D1) to the first time of disease progression. The primary analysis is based on the clinical benefit rate which is calculated as proportion of participants with a clinical benefit response relative to total number of response evaluable participants. Per RECIST v1.1 for target lesions: CR defined as disappearance of all target lesions; PR defined as >=30% decrease in the sum of the longest diameter of target lesions; SD does not qualify for CR, PR or Progression. All target lesions must be assessed. SD can follow PR only in the rare case that the sum increases by less than 20% from the nadir, but enough that a previously documented 30% decrease no longer holds. A Clopper-Pearson exact 95% CI for the clinical benefit rate is presented in the below table.
Time Frame: 16 weeks from Cycle 1 Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PF-05212384 (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants were given PF-05212384 QW (Days 1, 8, 15 and 22 of each cycle), with a ±3 day window.
- PF-05212384 (PI3K Activated): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K activated). Participants were given PF-05212384 QW (Days 1, 8, 15 and 22 of each cycle), with a ±3 day window.
- PF-05212384 (PI3K Basal + Activated): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal + activated). Participants were given PF-05212384 QW (Days 1, 8, 15 and 22 of each cycle), with a ±3 day window.
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 10 | 5 | 15
Percentage of participants | 52.6 [28.9 to 75.6] | 26.3 [9.1 to 51.2] | 39.5 [24.0 to 56.6]

3. Secondary Outcome: Objective Response for PF-04691502
Description: Objective response is defined as CR or PR. CR: Complete response: 2 or more objective statuses of CR a minimum of 4 weeks apart documented before PD. Partial response: 2 or more objective statuses of PR or better a minimum of 4 weeks apart documented before PD, but not qualifying as CR. Per RECIST v1.1 for target lesions: CR defined as disappearance of all target lesions; PR defined as >=30% decrease in the sum of the longest diameter of target lesions. The outcome data table below presents the number of participants with objective response as "yes" or "no". On 09 Oct 2012, Pfizer decided to stop enrollment into PF-04691502. While tumor assessment for PF-04691502 was included as a listing in the final report, formal efficacy analysis for PF-04691502 was not performed.
Time Frame: Randomization to objective progression, death or last tumor assessment without progression (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Participants response
Arm/Group | PF-04691502 (PI3K Basal) | PF-04691502 (PI3K Activated)
Number analyzed (Participants) | 4 | 11
Participants response
  Participants with "Yes" response | 0 | 0
  Participants with "No" response | 4 | 11

4. Secondary Outcome: Percentage of Participants With Objective Response for PF-05212384
Description: Objective response is defined as CR or PR. CR: Complete response: 2 or more objective statuses of CR a minimum of 4 weeks apart documented before PD. Partial response: 2 or more objective statuses of PR or better a minimum of 4 weeks apart documented before PD, but not qualifying as CR. Per RECIST v1.1 for target lesions: CR defined as disappearance of all target lesions; PR defined as >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Randomization to objective progression, death or last tumor assessment without progression (up to 12 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 19 | 19 | 38
Percentage of participants | 21.1 [6.1 to 45.6] | 15.8 [3.4 to 39.6] | 18.4 [7.7 to 34.3]

5. Secondary Outcome: Progression Free Survival for PF-04691502
Description: PFS is defined as the time from the date of cycle 1 day 1 to the date that objective progressive disease is documented or death due to any cause, whichever occurs first. PFS was characterized in terms of the median. Approximate 95% confidence interval corresponding to this estimate was computed. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions with a minimum absolute increase of 5 mm, or an unequivocal progression of non-target lesion, or the appearance of new lesions. On 09 Oct 2012, Pfizer decided to stop enrollment into PF-04691502. While tumor assessment for PF-04691502 was included as a listing in the final report, formal efficacy analysis for PF-04691502 was not performed.
Time Frame: From Cycle 1 Day 1 to objective progressive disease or death due to any cause whichever occurs first (up to 12 months)
Population: as for outcome 1
Measure: Number; unit: Time to Event (Days)
Arm/Group | PF-04691502 (PI3K Basal) | PF-04691502 (PI3K Activated)
Number analyzed (Participants) | 4 | 11
Time to Event (Days)
  Participant 1 | 1 | 0
  Participant 2 | 108 | 0
  Participant 3 | 50 | 0
  Participant 4 | 199 | 0
  Participant 5 | 0 | 54
  Participant 6 | 0 | 55
  Participant 7 | 0 | 51
  Participant 8 | 0 | 1
  Participant 9 | 0 | 54
  Participant 10 | 0 | 62
  Participant 11 | 0 | 53
  Participant 12 | 0 | 105
  Participant 13 | 0 | 1
  Participant 14 | 0 | 54
  Participant 15 | 0 | 54

6. Secondary Outcome: Progression Free Survival for PF-05212384
Description: PFS is defined as the time from the date of cycle 1 day 1 to the date that objective progressive disease is documented or death due to any cause, whichever occurs first. PFS was characterized in terms of the median. Approximate 95% confidence interval corresponding to this estimate was computed. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions with a minimum absolute increase of 5 mm, or an unequivocal progression of non-target lesion, or the appearance of new lesions.
Time Frame: From Cycle 1 Day 1 to objective progressive disease or death due to any cause whichever occurs first (up to 12 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 19 | 19 | 38
Days | 112.0 [59.0 to 167.0] | 89.0 [56.0 to 172.0] | 108.0 [62.0 to 149.0]

7. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 6 Months for PF-05212384
Description: Progression free survival is defined as the time from the date of cycle 1 day 1 to the date that objective progressive disease is documented or death due to any cause, whichever occurs first. PFS was characterized in terms of the probability of remaining progression-free at 6 months (based on Kaplan-Meier estimates). Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions with a minimum absolute increase of 5 mm, or an unequivocal progression of non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 19 | 19 | 38
Percentage of participants | 23.2 [7.3 to 44.1] | 25.0 [7.8 to 47.2] | 24.3 [11.6 to 39.5]

8. Secondary Outcome: Overall Survival (OS) for PF-05212384
Description: OS is defined as the time from the date of Cycle 1 Day 1 to the date of death.
Time Frame: 12 months
Population: Survival analysis was not performed as the study was terminated early. No data are available because data were not collected. The LIC reporting arm were not a part of the per protocol analysis set for summarizing response.
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Level of Each Pharmacodynamic Parameter at Specified Timepoints- Glucose (mg/dL)
Description: PD biomarkers are measured at screening (baseline) and multiple time points post baseline. Baseline is defined as the last measurement prior to dosing, which is the measurement at screening or the cycle 1 day 1 pre-dose measurement if collected. This outcome measure will be updated once the data is available with the supplemental clinical study report.
Time Frame: Baseline (Day -3) and Cycle1 to Cycle 5 where each cycle consist of 28 days
Population: Participants were analyzed on PD analysis set which consisted of all enrolled patients who started treatment and had a baseline as well as at least one post-baseline measurement for at least one PD biomarker. The PD biomarkers include serum glucose, insulin, HbA1c, cholesterol, and triglycerides.
Measure: Mean (Standard Deviation); unit: Glucose (mg/dL)
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 18 | 18 | 36
Glucose (mg/dL)
  Baseline | 98.5 (12.76) | 101.7 (26.56) | 100.1 (20.60)
  Cycle 1 Day 15 (n=18,17,35) | 105.3 (18.44) | 117.2 (61.04) | 111.1 (44.26)
  Cycle 1 Day 22 (n=2,1,3) | 103.0 (16.34) | 120.1 (0) | 108.7 (15.19)
  Cycle 2 Day 1 (n=17,14,31) | 103.7 (19.31) | 114.0 (39.42) | 108.3 (29.99)
  Cycle 2 Day 15 (n=17,8,25) | 104.8 (13.94) | 106.4 (19.36) | 105.3 (15.47)
  Cycle 3 Day 1 (n=14,10,24) | 100.6 (16.29) | 125.9 (74.50) | 111.1 (49.85)
  Cycle 4 Day 1 (n=12,7,19) | 96.3 (10.40) | 98.9 (10.20) | 97.3 (10.12)
  Cycle 5 Day 1 (n=9,4,13) | 103.2 (15.17) | 112.2 (24.37) | 106.0 (17.90)

10. Secondary Outcome: Level of Each Pharmacodynamic Parameter at Specified Timepoints- Insulin (UIU/mL)
Description: as for outcome 9
Time Frame: Baseline (Day -3) and Cycle1 to Cycle 5 where each cycle consist of 28 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Insulin (UIU/mL)
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 17 | 14 | 31
Insulin (UIU/mL)
  Baseline | 15.2 (12.68) | 14.4 (7.03) | 14.8 (10.36)
  Cycle 1 Day 15 (n=16,12,28) | 23.6 (14.69) | 35.9 (37.05) | 28.9 (26.79)
  Cycle 1 Day 22 (n=2,1,3) | 57.6 (51.18) | 29.1 (0) | 48.1 (39.75)
  Cycle 2 Day 1 (n=17,10,27) | 30.3 (28.92) | 28.9 (27.85) | 29.8 (27.99)
  Cycle 2 Day 15 (n=14,6,20) | 28.2 (29.56) | 21.9 (10.49) | 26.3 (25.21)
  Cycle 3 Day 1 (n=13,9,22) | 20.7 (13.65) | 35.1 (38.66) | 26.6 (26.99)
  Cycle 4 Day 1 (n=11,6,17) | 17.1 (10.04) | 24.8 (32.32) | 19.8 (20.10)
  Cycle 5 Day 1 (n=7,4,11) | 17.0 (15.56) | 15.7 (6.20) | 16.5 (12.54)

11. Secondary Outcome: Level of Each Pharmacodynamic Parameter at Specified Timepoints- Glycosylated Hemoglobin (HbA1c)
Description: as for outcome 9
Time Frame: Baseline (Day -3) and Cycle1 to Cycle 5 where each cycle consist of 28 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: HbA1c (mg/dL)
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 18 | 18 | 36
HbA1c (mg/dL)
  Baseline (n=15,14,29) | 7.8 (8.58) | 7.5 (6.15) | 7.7 (7.37)
  Cycle 1 Day 15 (n=4,2,6) | 14.7 (19.00) | 7.1 (1.34) | 12.2 (15.25)
  Cycle 2 Day 1 (n=15,13,28) | 8.4 (9.66) | 6.7 (1.16) | 7.6 (7.05)
  Cycle 2 Day 15 (n=3,0,3) | 6.7 (0.71) | NA (NA) — None of the participants were analyzed for arm PF-05212384 (PI3K activated) and hence data is not available. | 6.7 (0.71)
  Cycle 3 Day 1 (n=10,4,14) | 6.0 (0.78) | 7.3 (1.70) | 6.4 (1.19)
  Cycle 4 Day 1 (n=12,7,19) | 8.9 (10.13) | 6.9 (1.05) | 8.2 (8.01)
  Cycle 5 Day 1 (n=8,2,10) | 5.9 (0.89) | 31.5 (36.06) | 11.0 (16.17)

12. Secondary Outcome: Level of Each Pharmacodynamic Parameter at Specified Timepoints- Cholesterol (mg/dL)
Description: as for outcome 9
Time Frame: Baseline (Day -3) and Cycle1 to Cycle 3 where each cycle consist of 28 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Cholesterol (mg/dL)
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 18 | 18 | 36
Cholesterol (mg/dL)
  Baseline (n=11,4,15) | 213 (54.48) | 186.5 (52.43) | 205.9 (53.45)
  Cycle 1 Day 28 (n=15,7,22) | 214.9 (49.15) | 161.6 (86.51) | 198.0 (66.28)
  Cycle 2 Day 28 (n=16,6,22) | 229.8 (44.31) | 127.9 (108.69) | 202.0 (79.83)
  Cycle 3 Day 28 (n=11,4,15) | 230.5 (48.63) | 137.6 (107.02) | 205.7 (77.15)

13. Secondary Outcome: Level of Each Pharmacodynamic Parameter at Specified Timepoints- Triglycerides (mg/dL)
Description: as for outcome 9
Time Frame: Baseline (Day -3) and Cycle1 to Cycle 3 where each cycle consist of 28 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Triglycerides (mg/dL)
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 18 | 18 | 36
Triglycerides (mg/dL)
  Baseline (n=11,4,15) | 104.2 (40.95) | 133.4 (25.75) | 112.0 (38.96)
  Cycle 1 Day 28 (n=15,7,22) | 136.9 (70.03) | 134.5 (57.21) | 136.1 (64.85)
  Cycle 2 Day 28 (n=16,6,22) | 133.2 (71.40) | 117.1 (62.77) | 128.8 (68.07)
  Cycle 3 Day 28 (n=10,4,14) | 119.9 (64.22) | 130.4 (58.01) | 122.9 (60.47)

14. Secondary Outcome: Stathmin H Score [Mean (SD)] for Each Treatment Arm With Gene and/or Protein Expression Biomarkers in Biopsied Tumor Tissue
Description: Gene and/or protein expression biomarkers in biopsied tumor tissue relating to PI3K and/or mTOR pathway activation, such as PIK3CA and PIK3R1 mutations, PTEN protein levels, and PIK3CA gene amplification were to be assessed.
  Each slide was imaged by whole slide scanning and patient samples were scored as follows:
  * Pathologist manual score (0, 1+, 2+, 3+) for overall staining intensity of tumor tissue.
  * Percentage of positive tumor cells staining at 0, 1+, 2+, and 3+.
  * H-score value (integer between 0 and 300) for tumor cell staining was calculated. The higher the stathmin staining, the higher the stathmin H-score.
Time Frame: Prior to Cycle 1 Day 1
Population: Participants were analyzed as the molecular profiling tumor analysis set was defined as all enrolled patients who started treatment and had baseline tumor tissues (archived paraffin block or unstained slides or fresh tumor tissue sample) successfully analyzed for at least one of the biomarkers.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 21 | 19 | 40
Score | 96.4 (33.76) | 201.3 (34.87) | 146.2 (62.9)

15. Secondary Outcome: Percentage of Participants in Each Treatment Arm With Gene and/or Protein Expression Biomarkers- PIK3CA Amplification, KRAS Mutation P/N, KRAS Mutation OBSV, PTEN Stroma Manual Score, PTEN Tumor Manual Score, KRAS SCC and Stathmin H/L,Tissue.
Description: Gene and/or protein expression biomarkers in biopsied tumor tissue relating to PI3K and/or mTOR pathway activation, such as PIK3CA and PIK3R1 mutations, Phosphatase And Tensin Homolog (PTEN) protein levels, and PIK3CA gene amplification were to be assessed.
  Stained tissues were evaluated by a board-certified pathologist who provided a manual pathology score (i.e., 0, 1+, 2+, or 3+) and, if appropriate, comments upon the staining of the specimen.
  The directionality increases from 0 to 3+ with 0 being no staining for PTEN by IHC and 3+ being high staining intensity for PTEN.
Time Frame: Baseline and Cycle1 to Cycle 5 where each cycle consist of 28 days
Population: as for outcome 14
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 21 | 19 | 40
Percentage of participants
  PIK3CA Amplification, Amplified (n=17,15,32) | 5.9 (33.76) | 6.7 (34.87) | 6.3 (62.9)
  PIK3CA Amplification, Nonamplified (n=17,15,32) | 94.1 | 93.3 | 93.8
  KRAS Mutation, Positive (n=21,18,39) | 19.0 | 5.6 | 12.8
  KRAS Mutation, Negative (n=21,18,39) | 81.0 | 94.4 | 87.2
  KRAS Mutation OBSV, Gly12Asp (n=4,1,5) | 25.0 | 100 | 40.0
  KRAS Mutation OBSV, Gly12Cys (n=4,1,5) | 25.0 | 0 | 20.0
  KRAS Mutation OBSV, Gly12Val (n=4,1,5) | 50.0 | 0 | 40.0
  PTEN Stroma Manual Score, 1+ (n=21,19,40) | 4.8 | 0 | 2.5
  PTEN Stroma Manual Score, 2+ (n=21,19,40) | 28.6 | 26.3 | 27.5
  PTEN Stroma Manual Score, 3+ (n=21,19,40) | 66.7 | 73.7 | 70.0
  PTEN Tumor Manual Score, 0 (n=21,19,40) | 23.8 | 21.1 | 22.5
  PTEN Tumor Manual Score, 1+ (n=21,19,40) | 38.1 | 31.6 | 35.0
  PTEN Tumor Manual Score, 2+ (n=21,19,40) | 38.1 | 47.4 | 42.5
  KRAS SCC, Acceptable (n=21,18,39) | 100 | 100 | 100
  Stathmin H/L,Tissue, High (n=21,19,40) | 0 | 100 | 47.5
  Stathmin H/L,Tissue, Low (n=21,19,40) | 100 | 0 | 52.5

16. Secondary Outcome: Area Under the Serum Concentration Time Profile From Time Zero Extrapolated to Infinity (AUCinf) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours at Day 1
Population: Participants were analyzed on PK parameter analysis set which was defined as all treated patients who had at least one of the PK parameters of interest estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
ng.hr/mL | 15280 (24) | 14870 (40)

17. Secondary Outcome: Area Under the Serum Concentration Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours at Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/mL
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
ng.hr/mL | 15080 (24) | 15890 (52)

18. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours at Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
ng/mL | 9078 (36) | 7057 (84)

19. Secondary Outcome: Terminal Elimination Half Life (t½) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours at Day 1
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
hours | 35.02 (5.32) | 34.09 (8.87)

20. Secondary Outcome: Time for Cmax (Tmax) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours at Day 1
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
hours | 0.525 [0.500 to 1.07] | 0.650 [0.500 to 1.08]

21. Secondary Outcome: Clearance (CL) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours at Day 1
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
L/hr | 10.09 (24) | 10.36 (40)

22. Secondary Outcome: Steady State Volume of Distribution (Vss) of PF-05212384 at Each Specified Time Points.
Time Frame: Pre-dose: 0 hours, and Post dose: 0.5 (after end of infusion), 1, 2, 4, 6, 24, 72, and 120 hours
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated)
Number analyzed (Participants) | 19 | 15
Litres | 165.6 (32) | 174.9 (57)

23. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) - All Causalities
Description: Safety of participants in terms of TEAEs. Note: One subject treated with PF-05212384 had the stathmin status changed after randomization and was categorized under the corresponding arm.
Time Frame: From baseline (-3 days) until 35 days post last dose
Population: Participants were analyzed on safety analysis set which was defined as all enrolled patients who started treatment.
Measure: Number; unit: Number of AEs
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 20 | 20 | 40
Number of AEs | 244 | 269 | 513

24. Secondary Outcome: Summary of Treatment-emergent Adverse Events (TEAEs) - All Causalities
Description: as for outcome 23
Time Frame: From baseline (-3 days) until 35 days post last dose
Population: Participants were analyzed on safety analysis set which was defined as all enrolled patients who started treatment.
Measure: Number; unit: Number of participants
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 20 | 20 | 40
Number of participants
  Participants with AEs | 21 | 18 | 39
  Participants with Serious Adverse Events (SAEs) | 3 | 10 | 13
  Participants with Grade 3 or Grade 4 AEs | 7 | 14 | 21
  Participants with Grade 5 AEs | 1 | 1 | 2
  Permanently Discontinued due to AEs | 1 | 5 | 6
  Dose Reduced due to AEs | 1 | 5 | 6
  Temporary Discontinuations due to AEs | 8 | 10 | 16

25. Secondary Outcome: Number of Treatment-related TEAEs
Description: Safety of subject in terms of number of participants with treatment related AEs.
  Note: One subject treated with PF-05212384 had the stathmin status changed after randomization and was categorized under the corresponding arm.
Time Frame: From baseline (-3 days) until 35 days post last dose
Population: Participants were analyzed on safety analysis set which was defined as all enrolled patients who started treatment.
Measure: Number; unit: Number of AEs
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 20 | 20 | 40
Number of AEs | 158 | 161 | 319

26. Secondary Outcome: Summary of Treatment-related TEAEs
Description: as for outcome 25
Time Frame: From baseline (-3 days) until 35 days post last dose
Population: Participants were analyzed on safety analysis set which was defined as all enrolled patients who started treatment.
Measure: Number; unit: Number of participants
Arm/Group | PF-05212384 (PI3K Basal) | PF-05212384 (PI3K Activated) | PF-05212384 (PI3K Basal + Activated)
Number analyzed (Participants) | 20 | 20 | 3
Number of participants
  Participants with AEs | 21 | 18 | 39
  Participants with SAEs | 0 | 3 | 3
  Participants with Grade 3 or Grade 4 AEs | 4 | 9 | 13
  Participants with Grade 5 AEs | 0 | 0 | 0
  Permanently Discontinued due to AEs | 1 | 2 | 3
  Dose Reduced due to AEs | 1 | 4 | 5
  Temporary Discontinuations due to AEs | 6 | 7 | 13

ADVERSE EVENTS:
Time Frame: Maximum of treatment duration (i.e., 21 to 169 days for the PF 04691502 [PI3K basal and activated], 29 to 345 days for PF 05212384 PI3K basal and 1 to 400 days for PF 05212384 PI3K activated) + 28 days across all participants.
Description: There are inconsistency with the number of paticipants per arm in 'Participant flow section' and 'AE section' (both tables). This was because one participant treated with PF-05212384 and two subjects treated with PF-04691502 had their stathmin status changed after randomization and are categorized under the corresponding arm.
Groups:
- PF-05212384 154 mg (PI3K Basal): Eligible participants were categorized by PI3K pathway activation status (i.e. PI3K basal). Participants received PF-05212384 154 mg by 30 minute infusion at the study site, QW (Quaque [Once Weekly]) until they experienced unacceptable toxicity, disease progression, significant deviation, withdrawal of consent or death.
Arm/Group | PF-04691502 8 mg (PI3K Basal) | PF-04691502 6 mg (PI3K Basal) | PF-04691502 8 mg (PI3K Activated) | PF-04691502 6 mg (PI3K Activated) | PF-05212384 154 mg (PI3K Basal) | PF-05212384 154 mg (PI3K Activated) | Lead-in-cohort (LIC) PF-04691502 (4 mg) | LIC PF-05212384 (89 mg) | LIC PF-05212384 (154 mg)
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/1 | 7/9 | 1/3 | 3/21 | 10/19 | 1/3 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1 | 9/9 | 3/3 | 21/21 | 18/19 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502 8 mg (PI3K Basal) (N=5) | PF-04691502 6 mg (PI3K Basal) (N=1) | PF-04691502 8 mg (PI3K Activated) (N=9) | PF-04691502 6 mg (PI3K Activated) (N=3) | PF-05212384 154 mg (PI3K Basal) (N=21) | PF-05212384 154 mg (PI3K Activated) (N=19) | Lead-in-cohort (LIC) PF-04691502 (4 mg) (N=3) | LIC PF-05212384 (89 mg) (N=3) | LIC PF-05212384 (154 mg) (N=3)
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04691502 8 mg (PI3K Basal) (N=5) | PF-04691502 6 mg (PI3K Basal) (N=1) | PF-04691502 8 mg (PI3K Activated) (N=9) | PF-04691502 6 mg (PI3K Activated) (N=3) | PF-05212384 154 mg (PI3K Basal) (N=21) | PF-05212384 154 mg (PI3K Activated) (N=19) | Lead-in-cohort (LIC) PF-04691502 (4 mg) (N=3) | LIC PF-05212384 (89 mg) (N=3) | LIC PF-05212384 (154 mg) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
External Ear Inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Abnormal Sensation In Eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid Bleeding (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 4 | 0 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 7 | 6 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 7 | 2 | 8 | 10 | 1 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3 | 4 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | 5 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 5 | 1 | 12 | 10 | 1 | 3 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral Dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 5 | 3 | 1 | 3 | 3
Tooth Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 7 | 7 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 3 | 0 | 7 | 2 | 0 | 0 | 0
Catheter Site Bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter Site Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 6 | 2 | 5 | 10 | 1 | 0 | 1
Gait Disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion Site Extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion Site Rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 2
Medical Device Complication (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal Dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 2 | 0 | 3 | 1 | 12 | 8 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 1 | 0 | 2 | 5 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Genital Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 3 | 5 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood Alkaline Phosphatase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood Creatinine (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Magnesium Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Pressure Diastolic Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest X-Ray Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Glycosylated Haemoglobin Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0 | 0 | 3 | 3 | 2 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 6 | 1 | 9 | 8 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 7 | 0 | 4 | 3 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 0 | 1 | 2 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 1 | 3 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oncologic Complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 1 | 6 | 8 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dysthymic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 7 | 3 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 3 | 3 | 1 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hangnail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 6 | 3 | 3 | 1 | 2
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 5 | 0 | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dry Eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Noninfective Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.